CLINICAL TRIAL: NCT07164898
Title: Impact to Skin Due to Wet Pad Application. Skin Status and Change in the Stratum Corneum as Measured With 4 Instruments in an Elderly Population.
Brief Title: How Wet Pads Affect Elderly Skin: Measuring Changes in the Skin Barrier
Acronym: DROPBOX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Essity Hygiene and Health AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C3197
Record Dates: First submitted 2025-08-15; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Incontinence-associated Dermatitis
Keywords: "skin barrier" "absorbing incontinence product" elderly

STUDY DESIGN:
Intervention Model Description: Healthy volunteers get dry or wet test patches applied to the skin of the forearms. The cut outs are either dry or wetted with saline to 50% or 100% capacity. In total two pads are applied per forearm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Test patches (Experimental): Application of test patches. Each subject wear both low pH formula patches (intervention) and control patches without formula.
  Interventions: Device: Test patches

INTERVENTIONS:
Device: Test patches — Patches (incontinence product cut outs) either dry, 50% saturated with water or 100% saturated with water applied to the forearm and worn for 2 hours

SUMMARY:
The main aim of this study is to describe the effects of dry or wet incontinence pad material on the skin barrier function by measuring the changes of the stratum corneum on healthy participants due to the application of pads with varying wetness level to the forearm. Study findings have relevance for product development of absorbing incontinence products to further protect the skin from the damaging effects of excess moisture. Participants are subject to baseline measures of TEWL, SH, pH and water profile. Dry or wet pads are then added to the forearm skin and worn for two hours. After a recovery period, the SSWL, SH and water profile is measured. The study is conducted over a single 4h visit. As this is an explorative study no hypothesis is intended to be tested.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 65 years.
2. Mentally and physically able to participate in this study.
3. Written informed consent to participate in this study.
4. Intact skin on the volar forearms without skin irritation.

Exclusion Criteria:

1. Have any known allergies or intolerances to one or several components of the absorbing incontinence product.
2. Suffer from excessive sweating, hyperhidrosis.
3. Have any other condition that makes participation in the clinical investigation inappropriate, as judged by investigator.
4. Not be of childbearing potential.
5. Have an alcohol and/or drug dependency.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Trans Epidermal Water loss (TEWL) | 2 hours
  TEWL is measured at baseline and then after 2h of dry patch use the unit is g/m2*h. For the wet patches the follow up measurement is on skin surface water loss (SSWL) as the skin is not dry the unit is the same as for TEWL.

SECONDARY OUTCOMES:
Change in skin hydration | 2 hours
  Skin hydration (SH) as measured with moisture meter instrument under the test and control patches. Measure in arbitrary units (a.u).
Change in skin surface pH | 2 hours
  The pH change under the dry/wet patches are measured and compared.
Change skin water profile | 2 hours
  As measured Confocal raman microspectrometry. The water content (mass-% water) of skin at different depths is measured and compared for the skin under wet/dry patches.

CONTACTS AND LOCATIONS:
Overall Officials: Shabira Abbas, PhD, Principal Investigator — Essity Hygiene & Health AB
Locations (1):
- Essity Study Site, Mölndal, Sweden

IPD SHARING:
Plan to Share IPD: No